CLINICAL TRIAL: NCT03121612
Title: Randomised Trial Comparing CPAP Machines With Reusable vs Disposable Circuits
Brief Title: Comparison of CPAP Machines With Reusable vs Disposable Circuits
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient number of subjects
Sponsor: Medical Technology Transfer and Services Hong Kong Ltd (Industry)
Collaborators: MS Ramaiah Medical College & Hospitals (Other); Wellcome Trust (Other)
Responsible Party: Principal Investigator, Dr. Pradeep GCM, Neonatal Intensive Care Unit, MS Ramaiah Medical College & Hospitals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MTTS-01-2017
Record Dates: First submitted 2017-02-12; First posted 2017-04-20 (Actual); Results first posted 2019-11-04 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Respiratory Distress Syndrome, Newborn
Keywords: RDS
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn

STUDY DESIGN:
Masking Description: As the machines are physically distinct, blinding of participants, care providers and investigators is not feasible. The assessment of most outcomes cannot therefore be blinded, with one exception: x-rays for neonates with suspected pneumothorax will be provided to a radiologist for independent verification; the radiologist will not be in the nursery and will therefore be blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dolphin CPAP (Experimental): CPAP machine with oxygen intake and an on-board air compressor, and integrated blender and humidifier, delivering heated humidified blended gases through a Fisher-Paykel nasal mask. [Also includes built-in Massimo pulse oximeter, though this is not used for this study, to prevent differential measurement error in SpO2 measurement]
  Interventions: Device: CPAP
- Fisher-Paykel CPAP (Active Comparator): Fisher-Paykel (F&P) CPAP machine with separate oxygen and medical air intakes, with third-party FP-compliant blender, and F&P blender, delivering heated humidified blended gases through a Fisher-Paykel nasal mask.
  Interventions: Device: CPAP

INTERVENTIONS:
Device: CPAP — CPAP therapy

SUMMARY:
The study aims to assess the basic functionality of a newly designed CPAP machine with reusable circuits to existing machines with disposable circuits, for treatment of newborn infants diagnosed with respiratory distress syndrome. The assessment will compare a comprehensive list of physiological parameters over the first 72 hours of treatment, and will also monitor rates of side effects and adverse events. The null hypothesis is that infants treated on the two categories of machine (reusable vs disposable) will not differ in relation to key physiological parameters by more than 0.63 standard deviations.

DETAILED DESCRIPTION:
One of the commonest sources of serious newborn morbidity and mortality is difficulty with breathing. When this occurs, three main types of supportive therapy are available to increase the provision of oxygen to cells: a) passive provision of oxygen-enriched gases (i.e., higher than the 21% O2 found in the earth's atmosphere) through tubes in the nostrils, or by putting a hood over the baby's head and enriching the gases under that hood; b) provision of room air or oxygen-enriched gasses under pressure, frequently performed using a method called continuous positive airway pressure [CPAP] therapy; and/or c) by using a machine that is able to breath on behalf of the baby, most commonly referred to as mechanical ventilation [MV].

Passive therapy is the least invasive method but is also of limited benefit, particularly for infants born preterm. CPAP is more effective than passive methods because continuous distending pressure to the lungs allows better oxygen exchange; however, the distending pressure increases the risk of damage to the lung. MV is the only method that can be used on babies without a neurological impulse to breath, but the mechanical breathing action can damage the lungs, and MV is usually provided through a tube inserted into the lungs which increases the risk of lung infection; MV machines are also significantly more expensive than CPAP machines.

In high resource settings, CPAP is now the preferred method of providing oxygen for infants where passive therapy is insufficient, because of the lower infection risk, lower risk of lung damage, and relative ease of clinical care. CPAP is increasingly recommended for low resource settings, but the CPAP machines used in high resource settings are too expensive for low resource settings due to high-priced consumables ($US50-200/baby), and are usually unusable in low resource settings because they require 'medical air' (clean air in a cylinder, or through a piped wall system) with which to blend 100% oxygen. Low cost 'indigenous' machines ('jury-rigged' by hospital staff) have also been developed, but these do not provide the heated, humidified and blended gasses, that are recommended for CPAP.

This study seeks to evaluate a novel CPAP machine that provides heated, humidified, blended gasses, in line with recommendations for high-resource settings, while massively reducing costs by including re-usable tube sets and humidifiers that can be autoclaved, and with an on-board air-compressor to allow use in a broader range of clinical settings. By reducing the cost per CPAP treatment, such a machine can dramatically increase the number of hospitals in low resource settings that can provide high quality CPAP treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Infants born at Ramaiah Medical College hospital ('inborn infants');
2. Infants born elsewhere, and admitted to Ramaiah Medical College hospital under 6 hours of age ("outborn infants");
3. Infants with a gestational age at birth (weeks +days) in the range ≥ 28+0 to ≤ 36+6;
4. Infants thought to have RDS (clinically diagnosed after onset of respiratory distress <6 hours of age, sometimes confirmed by X-ray showing homogenous bilateral opacity) who would routinely be provided CPAP therapy; and
5. Infants <24 hours old at the time of fulfilling other inclusion criteria.

Exclusion Criteria:

1. Infants with a 1-minute Apgar score <3 (as a marker of severe birth asphyxia);
2. Infants who received MV prior to randomisation;
3. Infants with suspected meconium aspiration syndrome will be excluded to avoid any imbalance in this condition across groups;
4. Infants clinically suspected to have another specified serious condition as their main disease process, diagnosed prior to randomisation, specifically: cardiac anomaly, other congenital malformation with respiratory sequelae, septicaemia, pulmonary haemorrhage, pneumothorax, meningitis, poor respiratory effort or recurrent apnoea, or brain haemorrhage (IVH Grades III or IV);
5. Infants who have an airway abnormality precluding the use of the standard CPAP interface proposed for this study (e.g., Pierre-Robin sequence, cleft lip or cleft palate) or who have a neuromuscular condition that interferes with respiration;
6. Any infant whose treating clinician believes should not be randomised due to some other condition, or for any other reason (reason to be documented).

Ages: 1 Minute to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: G CM Pradeep, MD, Principal Investigator — MS Ramaiah Medical College
Locations (1):
- M.S. Ramaiah Medical College, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were no wash-out or run-in procedures. No enrolled participant was excluded from the study before randomisation.
Groups:
- Dolphin Continuous Positive Airway Pressure: Continuous Positive Airway Pressure (CPAP) machine with oxygen intake and an on-board air compressor, and integrated blender and humidifier, delivering heated humidified blended gases through a Fisher-Paykel nasal mask. [Also includes built-in Massimo pulse oximeter, though this is not used for this study, to prevent differential measurement error in SpO2 measurement]
  CPAP: CPAP therapy
- Fisher-Paykel Continuous Positive Airway Pressure: Fisher-Paykel (F&P) Continuous Positive Airway Pressure (CPAP) machine with separate oxygen and medical air intakes, with third-party FP-compliant blender, and F&P blender, delivering heated humidified blended gases through a Fisher-Paykel nasal mask.
  CPAP: CPAP therapy
Period: Overall Study
Arm/Group | Dolphin Continuous Positive Airway Pressure | Fisher-Paykel Continuous Positive Airway Pressure
Started | 26 | 25
Completed | 26 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dolphin Continuous Positive Airway Pressure | Fisher-Paykel Continuous Positive Airway Pressure | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Customized [Median (Inter-Quartile Range); unit: Weeks]
  Gestational age | 31.86 [31.29 to 32.71] | 31.57 [30.14 to 32.86] | 31.71 [30.57 to 32.86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 18 | 16 | 34
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  India | 25 | 26 | 51
Birthweight [Mean (Standard Deviation); unit: Grams] | 1409 (311) | 1434 (417) | 1421 (363)
FiO2 at baseline [Median (Inter-Quartile Range); unit: Percentage of inspired oxygen] | 40 [40 to 50] | 40 [40 to 50] | 40 [40 to 50]
SpO2 at baseline [Median (Inter-Quartile Range); unit: Percentage capillary oxygen saturation] | 96 [95 to 98] | 97 [94 to 98] | 97 [94 to 98]
Respiratory rate at baseline [Median (Inter-Quartile Range); unit: Breaths/minute] | 42.5 [40 to 44] | 43 [40 to 46] | 43 [40 to 44]
pH at baseline [Median (Inter-Quartile Range); unit: pH] — Population: Only 31/51 infants had a blood gas at baseline
  pH
    number analyzed (Participants) | 19 | 12 | 31
    (all) | 7.29 [7.22 to 7.35] | 7.34 [7.28 to 7.38] | 7.29 [7.23 to 7.36]
Partial pressure of arterial oxygen at baseline [Median (Inter-Quartile Range); unit: Torr] — Population: Only 31/51 infants had a blood gas at baseline
  Torr
    number analyzed (Participants) | 19 | 12 | 31
    (all) | 115 [74 to 140] | 139 [50 to 176] | 115 [65 to 152]
Partial pressure of arterial carbon dioxide at baseline [Median (Inter-Quartile Range); unit: Torr] — Population: Only 31/51 infants had a blood gas at baseline
  Torr
    number analyzed (Participants) | 19 | 12 | 31
    (all) | 38.9 [27.8 to 45.9] | 27.5 [23.4 to 40.4] | 37.2 [24.9 to 44.0]

OUTCOME MEASURES:

1. Primary Outcome: FiO2
Description: Fraction of inspired oxygen (FiO2), measured as a change from baseline as shown on the two machines.
  Note. Outcome contaminated. An SpO2 target of 90-95% reflects currently recommended practice for neonates; when SpO2 exceeds the target, FiO2 should be reduced. The majority of readings were at SpO2 > 95%, so FiO2 for these SpO2 readings reflects oxygen provided, not oxygen required to achieve the recommended SpO2 target range (i.e., the FiO2 provided was excessive, by an unknown amount).
Time Frame: 6, 12, 24, 48 and 72 hours after treatment commencement
Population: Number missing at each time point:
  6 hrs: 1 Dolphin (failed), 0 FP
  12 hrs: 1 Dolphin (failed), 1 FP (recovered)
  24 hrs: 6 Dolphin (2 failed + 4 recovered), 4 FP (all recovered)
  48 hrs: 16 Dolphin (3 failed + 13 recovered), 11 FP (1 failed + 10 recovered)
  72 hrs: 21 Dolphin (3 failed + 18 recovered), 21 FP (1 failed + 20 recovered)
Measure: Median (Inter-Quartile Range); unit: Percentage of inspired oxygen
Arm/Group | Dolphin CPAP | Fisher-Paykel CPAP
Number analyzed (Participants) | 26 | 25
Percentage of inspired oxygen
  Change at 6 hours: number analyzed (Participants) | 25 | 25
  Change at 6 hours | 0 [-7 to 0] | 0 [0 to 0]
  Change at 12 hours: number analyzed (Participants) | 25 | 24
  Change at 12 hours | 0 [-10 to 0] | 0 [-17 to 0]
  Change at 24 hours: number analyzed (Participants) | 20 | 21
  Change at 24 hours | -10 [-17 to 0] | -15 [-20 to 0]
  Change at 48 hours: number analyzed (Participants) | 10 | 14
  Change at 48 hours | -14.5 [-20 to -10] | -12.5 [-20 to 0]
  Change at 72 hours: number analyzed (Participants) | 5 | 4
  Change at 72 hours | -10 [-19 to -5] | -7.5 [-14.5 to -2.5]
Statistical Analysis 1: Comparison: Dolphin CPAP vs Fisher-Paykel CPAP; Analysis restricted to change at 6 hours, as least affected by missing data. Distribution non-normal, so non-parametric test (Wilcoxon) used; Test type: Superiority — Power calculated based on 40 infants in each arm, permitting detection of a difference of 0.67 SD between the groups with power of 80% and alpha=0.05. Study recruitment was below anticipated (51/80) despite extending the planned period of recruitment; p = 0.65, van Elteren's extension to Wilcoxon — Threshold for superiority p<0.05; primary outcome, so not adjusted for multiple comparisons; van Elteren's extension used to control for stratification by gestation
Statistical Analysis 2: Comparison: Dolphin CPAP vs Fisher-Paykel CPAP; Planned sub-group analysis for infants born at 28-33 gestational weeks (n=41). No adjustment for multiple comparisons; Test type: Superiority; p = 0.64, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Dolphin CPAP vs Fisher-Paykel CPAP; Planned sub-group analysis for infants born at 34-36 gestational weeks (n=10). No adjustment for multiple comparisons; Test type: Superiority; p = 1.0, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: SpO2
Description: Oxygen saturation by pulse oximetry (SpO2), measured as a change from baseline
  Note. Outcome contaminated. An SpO2 target of 90-95% reflects currently recommended practice for neonates. The majority of readings were at SpO2 > 95%, above SpO2 target (90-95%).
Time Frame: 6, 12, 24, 48 and 72 hours after treatment commencement
Population: Number missing:
  6 hrs: 1 Dolphin (failed), 0 FP
  12 hrs: 1 Dolphin (failed), 1 FP (recovered)
  24 hrs: 6 Dolphin (2 failed + 4 recovered), 4 FP (all recovered)
  48 hrs: 16 Dolphin (3 failed + 13 recovered), 11 FP (1 failed + 10 recovered)
  72 hrs: 21 Dolphin (3 failed + 18 recovered), 21 FP (1 failed + 20 recovered)
Measure: Median (Inter-Quartile Range); unit: Percentage capillary oxygen saturation
Arm/Group | Dolphin CPAP | Fisher-Paykel CPAP
Number analyzed (Participants) | 26 | 25
Percentage capillary oxygen saturation
  Change at 6 hours: number analyzed (Participants) | 25 | 25
  Change at 6 hours | 2 [0 to 3] | 1 [0 to 3]
  Change at 12 hours: number analyzed (Participants) | 25 | 24
  Change at 12 hours | 2 [0 to 3] | 1 [-0.5 to 3.5]
  Change at 24 hours: number analyzed (Participants) | 20 | 21
  Change at 24 hours | 1 [-1 to 2.5] | 0 [-2 to 1]
  Change at 48 hours: number analyzed (Participants) | 10 | 14
  Change at 48 hours | 1 [-4 to 1] | -0.5 [-2 to 1]
  Change at 72 hours: number analyzed (Participants) | 5 | 4
  Change at 72 hours | -1 [-5 to 4] | -0.5 [-1 to 0]
Statistical Analysis 1: Comparison: Dolphin CPAP vs Fisher-Paykel CPAP; Analysis restricted to change at 6 hours, as least affected by missing data. Distribution not normal by visual examination, so non-parametric test (Wilcoxon) used; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.80, van Elteren's extension to Wilcoxon — Threshold for superiority p<0.05; not adjusted for multiple comparisons; van Elteren's extension used to control for stratification by gestation

3. Secondary Outcome: Respiratory Rate
Description: Respiratory rate (breaths/minute), measured as a change from baseline
Time Frame: 6, 12, 24, 48 and 72 hours after treatment commencement
Population: Number missing (and thus imputed):
  6 hrs: 1 Dolphin (failed), 0 FP
  12 hrs: 1 Dolphin (failed), 1 FP (recovered)
  24 hrs: 6 Dolphin (2 failed + 4 recovered), 4 FP (all recovered)
  48 hrs: 16 Dolphin (3 failed + 13 recovered), 11 FP (1 failed + 10 recovered)
  72 hrs: 21 Dolphin (3 failed + 18 recovered), 21 FP (1 failed + 20 recovered)
Measure: Median (Inter-Quartile Range); unit: Breaths per minute
Arm/Group | Dolphin CPAP | Fisher-Paykel CPAP
Number analyzed (Participants) | 26 | 25
Breaths per minute
  Change at 6 hours: number analyzed (Participants) | 25 | 25
  Change at 6 hours | -2 [-2 to 3] | 0 [-2 to 2]
  Change at 12 hours: number analyzed (Participants) | 25 | 24
  Change at 12 hours | 0 [-2 to 0] | 0 [-2 to 2]
  Change at 24 hours: number analyzed (Participants) | 20 | 21
  Change at 24 hours | -2 [-4 to 2] | 0 [-2 to 2]
  Change at 48 hours: number analyzed (Participants) | 10 | 14
  Change at 48 hours | -1 [-4 to 2] | 0 [-2 to 2]
  Change at 72 hours: number analyzed (Participants) | 5 | 4
  Change at 72 hours | 0 [-2 to 4] | 0 [-1 to 1]
Statistical Analysis 1: Comparison: Dolphin CPAP vs Fisher-Paykel CPAP; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.86, van Elteren's extension to Wilcoxon — Threshold for superiority p<0.05; not adjusted for multiple comparisons; van Elteren's extension used to control for stratification by gestation

4. Secondary Outcome: Arterial pH
Description: pH measured as a change from baseline (where measured)
Time Frame: 6, 12, 24, 48 and 72 hours after treatment commencement (where available)
Population: Only 31/51 infants had a baseline blood gas taken, and only 7 of these had a second or subsequent test, with five of them at 6 hours, two each at 12 and 24 hours and one each at 48 and 72 hours. No statistical testing performed.
Measure: Median (Inter-Quartile Range); unit: pH
Arm/Group | Dolphin CPAP | Fisher-Paykel CPAP
Number analyzed (Participants) | 3 | 4
pH
  Change at 6 hours: number analyzed (Participants) | 2 | 3
  Change at 6 hours | 0.135 [0.08 to 0.19] | 0.05 [0.00 to 0.53]
  Change at 12 hours: number analyzed (Participants) | 1 | 1
  Change at 12 hours | 0.19 [0.19 to 0.19] | 0.23 [0.23 to 0.23]
  Change at 24 hours: number analyzed (Participants) | 2 | 0
  Change at 24 hours | 0.015 [0.0 to 0.03] |
  Change at 48 hours: number analyzed (Participants) | 0 | 1
  Change at 48 hours |  | 0.01 [0.01 to 0.01]
  Change at 72 hours: number analyzed (Participants) | 0 | 1
  Change at 72 hours |  | -0.01 [-0.01 to -0.01]

5. Secondary Outcome: Partial Pressure of Arterial Oxygen (PaO2)
Description: PaO2 measured as a change from baseline (where measured)
Time Frame: 6, 12, 24, 48 and 72 hours after treatment commencement (where available)
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: Torr
Arm/Group | Dolphin Continuous Positive Airway Pressure | Fisher-Paykel Continuous Positive Airway Pressure
Number analyzed (Participants) | 3 | 4
Torr
  Change at 6 hours: number analyzed (Participants) | 2 | 3
  Change at 6 hours | -138 [-179 to -97] | -47 [-67 to 0]
  Change at 12 hours: number analyzed (Participants) | 1 | 1
  Change at 12 hours | -60.2 [-60.2 to -60.2] | 12.1 [12.1 to 12.1]
  Change at 24 hours: number analyzed (Participants) | 2 | 0
  Change at 24 hours | -42.5 [-85 to 0] |
  Change at 48 hours: number analyzed (Participants) | 0 | 1
  Change at 48 hours |  | -9.3 [-9.3 to -9.3]
  Change at 72 hours: number analyzed (Participants) | 0 | 1
  Change at 72 hours |  | 15.6 [15.6 to 15.6]

6. Secondary Outcome: Partial Pressure of Arterial Carbon Dioxide (PaCO2)
Description: PaCO2 measured as a change from baseline (where measured)
Time Frame: 6, 12, 24, 48 and 72 hours after treatment commencement (where available)
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: Torr
Arm/Group | Dolphin Continuous Positive Airway Pressure | Fisher-Paykel Continuous Positive Airway Pressure
Number analyzed (Participants) | 3 | 4
Torr
  Change at 6 hours: number analyzed (Participants) | 2 | 3
  Change at 6 hours | -17 [-27 to -7] | -9 [-30 to 0]
  Change at 12 hours: number analyzed (Participants) | 1 | 1
  Change at 12 hours | -18.6 [-18.6 to -18.6] | -5.9 [-5.9 to -5.9]
  Change at 24 hours: number analyzed (Participants) | 2 | 0
  Change at 24 hours | -12 [-24 to 0] |
  Change at 48 hours: number analyzed (Participants) | 0 | 1
  Change at 48 hours |  | -0.1 [-0.1 to -0.1]
  Change at 72 hours: number analyzed (Participants) | 0 | 1
  Change at 72 hours |  | 6.4 [6.4 to 6.4]

7. Secondary Outcome: Number of Participants Who Died or Needed Intubation and/or Mechanical Ventilation, as a Measure of CPAP Failure, Measured to Date and Time of Cessation of CPAP Treatment
Description: Death or need for intubation and mechanical ventilation as demonstrated by an FiO2 requirement ≥ 60% for ≥ 1 hour to maintain SpO2 at 90-95%
  Note. An SpO2 target of 90-95% reflects currently recommended practice for neonates. FiO2 and SpO2 at time of intubation and ventilation not separately recorded, so we report this endpoint as recorded by clinicians, assuming that they have verified FiO2 [≥ 60% for ≥ 1 hour] and SpO2 [targeting 90-95%] requirements at the time of intubation and ventilation. If SpO2 was actually >95% (not 90-95%) at the time of intubation and ventilation, then FiO2 would be higher than required to meet the target range, by an unknown amount (possibly not meeting the FiO2 threshold of ≥ 60% for ≥ 1 hour, required to justify intubation and ventilation). We note this potential source of contamination because the results of Outcome #2 show that the majority of SpO2 readings were >95%.
Time Frame: From date and time of randomization to date and time of cessation of CPAP treatment, or until date and time of hospital discharge, if infant is on CPAP treatment until discharged (i.e., dies or is transferred), assessed to a maximum of 2 months of age.
Measure: Count of Participants; unit: Participants
Arm/Group | Dolphin CPAP | Fisher-Paykel CPAP
Number analyzed (Participants) | 26 | 25
Participants | 3 | 2
Statistical Analysis 1: Comparison: Dolphin CPAP vs Fisher-Paykel CPAP; Test type: Superiority; p = 1.0, Fisher Exact — Not adjusted for multiple comparisons; No failures in older stratum, so stratification by gestational age-group not controlled for in analysis

8. Secondary Outcome: Surfactant Provided When FiO2 > 40% to Maintain SpO2 at 90-95% for ≥ 30 Minutes, With Respiratory Distress Syndrome Confirmed by Chest X-Ray
Description: Surfactant provided when FiO2 > 40% to maintain SpO2 at 90-95% for ≥ 30 minutes, with Respiratory Distress Syndrome confirmed by chest X-Ray
  Note that endpoint likely corrupted because SpO2 was not routinely targeting 90-95%, and large number of infants received surfactant before achieving >40% or without having x-ray confirmation of RDS.
Time Frame: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Dolphin CPAP | Fisher-Paykel CPAP
Number analyzed (Participants) | 26 | 25
Participants | 3 | 1
Statistical Analysis 1: Comparison: Dolphin CPAP vs Fisher-Paykel CPAP; Test type: Superiority; p = 0.33, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Controlling for stratification by gestational group

9. Secondary Outcome: CPAP Failure or Surfactant Provision
Description: Outcomes 6 or 7
  Note that endpoint likely corrupted because SpO2 was not routinely targeting 90-95%, and large number of infants received surfactant before achieving >40% or without having x-ray confirmation of RDS.
Time Frame: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Dolphin CPAP | Fisher-Paykel CPAP
Number analyzed (Participants) | 26 | 25
Participants | 6 | 3
Statistical Analysis 1: Comparison: Dolphin CPAP vs Fisher-Paykel CPAP; Test type: Superiority; p = 0.31, Cochran-Mantel-Haenszel — Not adjusted for multiple comparisons; Controlling for stratification by gestational age-group

10. Secondary Outcome: CPAP Duration
Description: Duration of CPAP treatment (hours) in infants that do not fail CPAP
Time Frame: as for outcome 7
Population: Excludes 3 Dolphin and 2 FP randomised infants that failed treatment (escalated to mechanical ventilation)
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Dolphin CPAP | Fisher-Paykel CPAP
Number analyzed (Participants) | 23 | 23
Hours | 46.9 [42.1 to 70.0] | 56.5 [38.0 to 65.0]
Statistical Analysis 1: Comparison: Dolphin CPAP vs Fisher-Paykel CPAP; Test type: Superiority; p = 0.81, van Elteren's extension to Wilcoxon — Not adjusted for multiple comparisons; van Elteren's extension used to control for stratification by gestation

11. Secondary Outcome: Serious Adverse Event
Description: A Serious adverse Event (SAEs) is any untoward medial occurrence that:
  * Results in death;
  * Is life-threatening; [NOTE: the term "life-threatening" in the definition of "serious" refers to an event in which the patient was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe.]
  * Requires inpatient hospitalisation or prolongation of existing hospitalisation;
  * Results in persistent or significant disability/incapacity, or
  * Is a congenital anomaly/birth defect
Time Frame: From date and time of birth to date and time of hospital discharge, assessed to a maximum of 2 months of age.
Population: The infant that died recovered after CPAP but was subsequently treated for apnea and a patent ductus arteriosus. Twelve days after CPAP cessation the infant commenced antibiotics for elevated CRP and was intubated and ventilated and died. The Data Safety Monitoring Committee determined that the death was unrelated to treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Dolphin CPAP | Fisher-Paykel CPAP
Number analyzed (Participants) | 26 | 25
Participants | 1 | 0
Statistical Analysis 1: Comparison: Dolphin CPAP vs Fisher-Paykel CPAP; Test type: Superiority; p = 1.0, Fisher Exact

12. Secondary Outcome: Sentinel Outcome #1
Description: Damage to the nasal septum
Time Frame: From date and time of randomization to date and time of CPAP cessation, assessed to a maximum of 2 months of age.
Measure: Count of Participants; unit: Participants
Arm/Group | Dolphin CPAP | Fisher-Paykel CPAP
Number analyzed (Participants) | 26 | 25
Participants | 0 | 0

13. Secondary Outcome: Sentinel Outcome #2
Description: Damage to the nares of the infant
Time Frame: From date and time of randomization to date and time of CPAP cessation, assessed to a maximum of 2 months of age.
Measure: Count of Participants; unit: Participants
Arm/Group | Dolphin CPAP | Fisher-Paykel CPAP
Number analyzed (Participants) | 26 | 25
Participants | 0 | 0

14. Secondary Outcome: Sentinel Outcome #3
Description: Pneumothorax as diagnosed by X-ray
Time Frame: From date and time of randomization to date and time of CPAP cessation, assessed to a maximum of 2 months of age.
Measure: Count of Participants; unit: Participants
Arm/Group | Dolphin CPAP | Fisher-Paykel CPAP
Number analyzed (Participants) | 26 | 25
Participants | 0 | 0

15. Secondary Outcome: Sentinel Outcome #4
Description: Intra-ventricular haemorrhage (IVH), intra-cranial haemorrhage (ICH), or periventricular leukomalacia (PVL) as diagnosed by cranial ultrasound scan
Time Frame: From date and time of randomization to date and time of CPAP cessation, assessed to a maximum of 2 months of age.
Measure: Count of Participants; unit: Participants
Arm/Group | Dolphin CPAP | Fisher-Paykel CPAP
Number analyzed (Participants) | 26 | 25
Participants | 0 | 0

16. Secondary Outcome: Sentinel Outcome #5
Description: FiO2 ≥ 60% to maintain SpO2 at 90-95% for one hour or more, during CPAP treatment
Time Frame: From date and time of randomization to date and time of CPAP cessation, assessed to a maximum of 2 months of age.
Measure: Count of Participants; unit: Participants
Arm/Group | Dolphin CPAP | Fisher-Paykel CPAP
Number analyzed (Participants) | 26 | 25
Participants | 0 | 0

17. Secondary Outcome: Sentinel Outcome #6
Description: Intubation and mechanical ventilation
  Note. An SpO2 target of 90-95% reflects currently recommended practice for neonates. FiO2 and SpO2 at time of intubation and ventilation not separately recorded, so we report this endpoint as recorded by clinicians, assuming that they have verified FiO2 [≥ 60% for ≥ 1 hour] and SpO2 [targeting 90-95%] requirements at the time of intubation and ventilation. If SpO2 was actually >95% (not 90-95%) at the time of intubation and ventilation, then FiO2 would be higher than required to meet the target range, by an unknown amount (possibly not meeting the FiO2 threshold of ≥ 60% for ≥ 1 hour, required to justify intubation and ventilation). We note this potential source of contamination because the results of Outcome #2 show that the majority of SpO2 readings were >95%.
Time Frame: From date and time of randomization to date and time of CPAP cessation, assessed to a maximum of 2 months of age.
Measure: Count of Participants; unit: Participants
Arm/Group | Dolphin CPAP | Fisher-Paykel CPAP
Number analyzed (Participants) | 26 | 25
Participants | 3 | 2
Statistical Analysis 1: Comparison: Dolphin CPAP vs Fisher-Paykel CPAP; Test type: Superiority; p = 1.0, Fisher Exact — No adjustment for multiple comparisons; No failures in older stratum, so stratification by gestational age-group not controlled for in analysis

18. Secondary Outcome: Sentinel Outcome #7
Description: For infants born at 28+0 to 33+6 weeks' gestation, oxygen dependent at 36 weeks' gestation
Time Frame: From date and time of randomization to date and time of CPAP cessation, assessed to a maximum of 2 months of age.
Measure: Count of Participants; unit: Participants
Arm/Group | Dolphin CPAP | Fisher-Paykel CPAP
Number analyzed (Participants) | 26 | 25
Participants | 0 | 0

19. Secondary Outcome: Sentinel Outcome #8
Description: Death of the infant before hospitals discharge
Time Frame: From date and time of randomization to date and time of hospital discharge, assessed to a maximum of 2 months of age.
Population: The infant that died recovered after CPAP but was subsequently treated for apnoeas and a patent ductus arteriosus. Twelve days after CPAP cessation the infant commenced antibiotics for elevated CRP and was intubated and ventilated and died. The Data Safety Monitoring Committee determined that the death was unrelated to treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Dolphin CPAP | Fisher-Paykel CPAP
Number analyzed (Participants) | 26 | 25
Participants | 1 | 0
Statistical Analysis 1: Comparison: Dolphin CPAP vs Fisher-Paykel CPAP; Test type: Superiority; p = 1.0, Fisher Exact; No adjustment for multiple comparisons

ADVERSE EVENTS:
Time Frame: Adverse event data were collected till hospital discharge or two months of age, whichever is earlier.
Description: One serious adverse events was monitored, death.
Arm/Group | Dolphin CPAP | Fisher-Paykel CPAP
All-Cause Mortality (participants affected / at risk) | 1/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/26 | 0/25
Other Adverse Events (participants affected / at risk) | 4/26 | 2/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dolphin CPAP (N=26) | Fisher-Paykel CPAP (N=25)
Death (Infections and infestations) | 1 (1) | 0 (0) — As required by the governing ethics committee, death for any reason before hospital discharge was defined as a serious adverse event. Details of the death are reported at Outcome #19.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dolphin CPAP (N=26) | Fisher-Paykel CPAP (N=25)
Intubation & Mechanical Ventilation (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) — Intubation and mechanical ventilation after FiO2>=60%
Culture confirmed infection (Infections and infestations) | 2 (2) | 1 (1) — Diagnosed with Klebsiella Pneumoniae

LIMITATIONS AND CAVEATS:
1. Sample size achieved (n=51) was fewer than than planned (n=80).
2. Many of the outcomes were affected by a failure to target SpO2 of 90-95% as anticipated in the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-08-31): https://cdn.clinicaltrials.gov/large-docs/12/NCT03121612/SAP_000.pdf
  • Study Protocol (2017-04-03): https://cdn.clinicaltrials.gov/large-docs/12/NCT03121612/Prot_001.pdf